CLINICAL TRIAL: NCT06824233
Title: Deciphering the Molecular Landscape of Diabetic Cardiovascular Complications Based on Multi-Omics Analysis
Brief Title: Diabetic Cardiovascular Complications: Multi-Omics Analysis
Acronym: D-CCMOA
Status: Not yet recruiting | Type: Observational
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: LYF20240324
Record Dates: First submitted 2025-02-07; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Diabetes
Keywords: Multi-Omics Analysis; Diabetes; Cardiovascular Complications
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The study will collect several types of biological samples from participants, but all samples will be destroyed immediately after testing. These include:
  Blood Samples (5 mL per participant): Blood samples will be collected for genomics, transcriptomics, and proteomics analysis. The blood will be processed to isolate plasma, serum, and peripheral blood mononuclear cells (PBMCs) for the following purposes:
  1. Genomic analysis
  2. Transcriptomic analysis
  3. Proteomic analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- No Diabetes or Cardiovascular Complications Group: This group consists of individuals who do not have diabetes or cardiovascular complications. They serve as a control group for comparison with the other cohorts. Participants in this group will undergo the same clinical assessments and provide biological samples for multi-omics analysis to identify molecular differences between individuals with and without T2DM and cardiovascular issues.
- T2DM without Cardiovascular Complications Group: This group includes individuals diagnosed with type 2 diabetes but without any cardiovascular complications at the time of enrollment. The goal is to explore the molecular effects of T2DM on biological networks independent of cardiovascular issues. Participants will provide blood samples for genomic, transcriptomic, and proteomic analysis and undergo standard clinical tests, including echocardiograms and measurements of vascular health.
- T2DM with Cardiovascular Complications Group: This group consists of T2DM patients who have developed cardiovascular complications, such as coronary artery disease or heart failure. This cohort will be studied to identify how cardiovascular complications further alter molecular networks in individuals with T2DM. Blood samples will be analyzed for genomics, gene expression, and protein profiles, and participants will undergo additional clinical assessments, including vascular imaging and ankle-brachial index measurements.

SUMMARY:
The goal of this observational study is to learn about the molecular mechanisms underlying cardiovascular complications in individuals with type 2 diabetes (T2DM) and how they differ from healthy individuals. The study will also identify biomarkers and potential therapeutic targets for better managing diabetes-related heart disease.

The main questions it aims to answer are:

1. What molecular changes are associated with cardiovascular complications in T2DM patients compared to healthy individuals?
2. How do genetic, gene expression, and protein profiles differ between T2DM patients with and without cardiovascular complications? Researchers will compare the molecular profiles of three groups: healthy controls, individuals with T2DM but no cardiovascular complications, and those with T2DM and cardiovascular complications.

Participants will:

1. Provide blood samples for genomics, transcriptomics, and proteomics analysis
2. Undergo standard clinical tests such as blood pressure, echocardiogram, and ankle-brachial index measurements
3. Be followed for 12 to 24 months to track the development of cardiovascular events Participate in follow-up phone interviews to record major cardiovascular events like heart attacks or strokes

ELIGIBILITY:
Inclusion Criteria:

1. Age: Patients aged between 20 and 70 years.
2. Coronary Angiography: Patients who have undergone coronary angiography at the Second Xiangya Hospital of Central South University for various reasons.
3. Informed Consent: Patients who have signed the informed consent form and are willing to participate in the collection and analysis of multi-omics data.
4. Medical History and Samples: Patients who can provide complete medical history and biological samples.

Exclusion Criteria:

1. Severe Diseases or Malignancy: Patients with other severe diseases or malignancies that may affect the study.
2. Cognitive or Psychiatric Disorders: Patients with cognitive or psychiatric disorders that would prevent participation or cooperation in the study.
3. Pregnancy or Lactation: Women who are pregnant or breastfeeding.
4. Short Life Expectancy: Patients with a life expectancy of less than 6 months.
5. Inability to Provide Consent: Patients unable or unwilling to provide informed consent.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients who have undergone coronary angiography at the Second Xiangya Hospital of Central South University for various reasons. The study will involve individuals aged between 20 and 70 years who meet the inclusion criteria, including providing informed consent and the ability to supply complete medical history and biological samples. The population will encompass individuals with varying levels of cardiovascular health, including those with and without cardiovascular complications, to enable comprehensive multi-omics analysis and long-term cardiovascular event tracking.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Major Adverse Cardiovascular Events (MACE) | From enrollment to the end of treatment at 12 months and 24 months
  Description: To assess the occurrence of major adverse cardiovascular events (MACE), including myocardial infarction, stroke, or heart failure, over the 2-year follow-up period.
  Time Frame: 12 months and 24 months follow-up. Measurement Method: Clinical assessments through medical records, including hospitalizations, laboratory data, echocardiograms, and imaging techniques (e.g., vascular imaging, ABI, carotid ultrasound).

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 3 months and ending 3 years after the publication of results
Access Criteria: To access the IPD and supporting information, interested parties should contact the principal investigator.